CLINICAL TRIAL: NCT05216627
Title: COVID SAFE 2.0: COVID-19 Screening Program
Brief Title: COVID-19 Screening Program
Acronym: COVID SAFE 2
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 850592
Record Dates: First submitted 2022-01-27; First posted 2022-01-31 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PSOM staff, trainees, or faculty who participate in the point of care testing: The cohort will be offered access to a self-administered saliva-based viral test is a small funnel and a tube in which participants will put their saliva into. When they are ready to self-collect their saliva sample, they will be instructed to not eat or drink for 30 minutes prior to collecting their saliva and to collect saliva in an isolated room. We will evaluate the implementation of this viral test.
  Interventions: Diagnostic Test: Self-administered saliva-based viral testing

INTERVENTIONS:
Diagnostic Test: Self-administered saliva-based viral testing — Participants will be instructed on how to inactivate the virus and bring their sample to their laboratory's central PCR machine, where they will take an assay test. They will be instructed to collect saliva into a 1.5 milliliter (mL) collection tube containing inactivation buffer (TCEP and EDTA) using a small funnel and inactivate at 95°C for 10 minutes. Participants will then transfer 6ul of saliva into 2 PCR tubes containing amplification master mix and primers, put tubes in a heat block or PCR machine at 65°C for 45 minutes and assess fluorescence using a simple battery-powered fluorescence viewer. Once they assess their sample, they will be instructed to dispose of the saliva sample safely and in accordance with best laboratory practices. No saliva samples will be collected by the research team at any time as part of this study.

SUMMARY:
In view of the recent COVID surge and difficulties in obtaining testing, we aim to increase Point of Care (POC) testing, whereby University of Pennsylvania (Penn) faculty, staff, and trainees who are working in person at Perelman School of Medicine (PSOM) laboratories can self-test. The purpose of this study is to evaluate the implementation of this POC testing program. We will not be collecting any samples as part of this study. This will ensure that individuals can rapidly identify if they have COVID-19 while balancing use, acceptability, appropriateness, and feasibility. We will start with a pilot phase whereby we will evaluate the implementation of a POC version of COVID-19 screening program that will coordinate several existing systems at the University of Pennsylvania including voluntary, self-administered saliva-based viral testing. We will pilot this program to a small cohort of PSOM labs and then test implementation of the self-testing of the POC version of COVID-19 screening across all PSOM labs for those who wish to participate. All results will be self-reported and will not be used to validate any tests or support any future approval from the FDA. No data from this study will go into the participants' Electronic Medical Record (EMR).

DETAILED DESCRIPTION:
Background: The coronavirus disease (COVID-19) pandemic has resulted in close to 300,000,000 reported cases worldwide, including more than 58,000,000 reported cases and 800,000 deaths in the United States [1,2]. Initial efforts to address the COVID-19 pandemic were aimed at testing symptomatic individuals, implementing stay-in-place orders, and at increasing hospital capacity to meet surge demands [3]. Currently, we are going through an unprecedented surge in the total number of cases - mostly due to the spread of the Omicron variant. While we continue to confront the current crisis, a complete lockdown as seen in 2020 is not desirable or being planned. We must address the current issue and also plan for the future by putting in place tools to enhance our ability to conduct effective screening, containment, and case management. Future variants may cause similar delays in testing availability.

Widespread COVID-19 testing is needed to safely and effectively operate schools, workplaces, and businesses across the US. However, currently approved clinical testing options require reagents that are limited in supply and expensive quantitative polymerase chain reaction (qPCR) machines, severely hindering scalability [4] coupled with acute shortage of person-power. In response to limited clinical testing options, rapid antigen tests that are available to purchase over-the-counter and can be self-administered have become recently a popular testing approach; however, these tests are expensive, in short supply, and may not be as sensitive in detecting Omicron variant compared to polymerase chain reaction (PCR) tests [5]. Emerging evidence indicates that saliva testing with the option of self-administration of testing can accurately identify COVID-19 viral infection [6]. Moreover, this approach provides an option for the easy, safe and convenient collection of samples required for testing without traveling to a doctor's office, hospital, or testing site. Point of care testing (i.e. using saliva-based self-collection to administer screening for COVID-19 in one's own laboratory setting) utilizes testing equipment that is readily available to our workforce, leverages their existing training, and benefits from existing institutional health and safety infrastructure.

Self-administration of saliva testing also reduces exposure of health care workers to the virus and preserves limited personal protective equipment [7]. Additional diagnostic testing options will continue to increase staff access.

For these reasons, we propose to evaluate the implementation of a COVID-19 POC screening program that uses saliva-based self-testing and to pilot test approaches to improve program enrollment.

Objective: The primary objective of the study is to evaluate the use, acceptability, appropriateness, and feasibility of implementing a voluntary COVID-19 Point of Care (POC) screening program with Penn faculty, staff, and trainees that uses saliva-based self-collection followed by testing in their own PSOM laboratories. A secondary objective is to learn about self-reported test results, program usability, user burden, participant experience, program ease, program continuation and availability. Another secondary objective is to learn about individual's perspectives about the program.

Study Design: This is an implementation clinical trial that we anticipate lasting up to two months. In the first phase, we will pilot the approach with four PSOM laboratories. We plan to enroll up to 50 people across these labs during the pilot phase. Labs will be located on Penn campus. We will pilot test the best manner to distribute saliva collection test kits and assay tests to participants and elicit rapid feedback for one week. We will apply feedback in real time to improve the distribution method. In the second phase, we will roll out the clinical trial more broadly across all interested PSOM laboratories. We anticipate enrolling up to 500 participants across all PSOM laboratories. All participants will be Penn employees (faculty, staff, and trainees) who work in a PSOM laboratory.

All participants will be required to provide informed consent and watch a training video before self-collecting their first saliva sample. All participants will be told they can collect saliva samples as much or as little as they want - but no more than daily for up to four weeks. They will also be asked to complete online surveys weekly for up to four weeks. These surveys are expected to take about 15 minutes to complete. See below for table of survey measures and frequency. A subset of participants will also be asked to participate in a one-time qualitative interview after the point of care testing program is over. This interview is expected to take about 30 minutes.

ELIGIBILITY:
To be eligible, participants must:

1. Be 18 years or older
2. Be University of Pennsylvania staff, faculty or trainee who is working in person on campus at a PSOM laboratory
3. Have knowledge of safe practices in and access to a biological safety cabinet
4. Have knowledge and access to pipet and PCR machine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PSOM staff, faculty, or trainees who work in person on campus in a PSOM laboratory
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rinad Beidas, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data (IPD) to other researchers

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PSOM Staff, Trainees, or Faculty Who Participate in the Point of Care Testing
Started | 61
Completed | 61
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PSOM Staff, Trainees, or Faculty Who Participate in the Point of Care Testing
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Some participants did not provide their age.
  years
    number analyzed (Participants) | 45
    (all) | 37.9 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 59
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 39
  More than one race | 2
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 61
Study Participation Level [Count of Participants; unit: Participants] — Participants came from 15 laboratories. Each laboratory had a captain responsible for tracking their lab's participation, collecting the necessary materials for their colleagues, and responding to outcome-related survey questions. Participants who were not captains participated in testing and did not answer outcome-related survey questions.
  Participants
    Lab Captains | 15
    Non-Captains | 46

OUTCOME MEASURES:

1. Primary Outcome: Use of a Voluntary COVID-19 Point of Care (POC) Screening Program
Description: How often they use the POC screening program
Time Frame: fourteen weeks
Population: Lab-wide screening test completion was reported to the study team by captains on behalf of participants from their respective labs. Fifteen captains participated over the course of the program.
Measure: Number; unit: total completed screening tests reported
Arm/Group | PSOM Staff, Trainees, or Faculty Who Participate in the Point of Care Testing
Number analyzed (Participants) | 15
total completed screening tests reported | 238

2. Primary Outcome: Acceptability of Implementing a Voluntary COVID-19 Point of Care (POC) Screening Program
Description: Self-reported acceptability of implementing POC screening program using the Acceptability of Intervention Measure (i.e., "Point of care testing is acceptable to me"). Scale values: 1 (completely disagree) to 5 (completely agree).
Time Frame: fourteen weeks
Population: Only the 15 lab captains completed surveys related to this outcome. As such, results for this outcome were only collected from the 15 lab captains, not all participants. Screening tests were conducted by the 15 lab captains on behalf of participants from their respective labs.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: survey responses
Arm/Group | PSOM Staff, Trainees, or Faculty Who Participate in the Point of Care Testing
Number analyzed (Participants) | 15
Number analyzed (survey responses) | 82
score on a scale | 4.36 (0.72)

3. Primary Outcome: Appropriateness of Implementing a Voluntary COVID-19 Point of Care (POC) Screening Program
Description: Self-reported appropriateness of implementing POC screening program using the Intervention Appropriateness Measure (i.e., "Point of care testing seems appropriate."). Scale values: 1 (completely disagree) to 5 (completely agree).
Time Frame: fourteen weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: survey responses
Arm/Group | PSOM Staff, Trainees, or Faculty Who Participate in the Point of Care Testing
Number analyzed (Participants) | 15
Number analyzed (survey responses) | 82
score on a scale | 4.40 (0.72)

4. Primary Outcome: Feasibility of Implementing a Voluntary COVID-19 Point of Care (POC) Screening Program
Description: Self-reported feasibility of implementing POC screening program using the Feasibility of Intervention Measure (i.e., "Point of care testing seems feasible."). Scale values: 1 (completely disagree) to 5 (completely agree).
Time Frame: fourteen weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: survey responses
Arm/Group | PSOM Staff, Trainees, or Faculty Who Participate in the Point of Care Testing
Number analyzed (Participants) | 15
Number analyzed (survey responses) | 82
score on a scale | 4.29 (0.75)

5. Secondary Outcome: Self Report of Test Results
Description: Self-report of if participant received any positive test results from saliva-based viral test or Clinical Laboratory Improvement Amendments (CLIA) approved test
Time Frame: four weeks
Population: Given participant preferences to retain privacy, individual counts of positive tests were not tracked and self-reports of test results were not collected. However, when completing the survey on their colleagues' behalf, lab captains could note whether anyone in their labs received a positive test result, and they also had the option not to disclose results. The count for this measure refers to the number of labs which reported a positive test result during the study period.
Measure: Number; unit: laboratories
Units Other Than Participants: survey responses
Arm/Group | PSOM Staff, Trainees, or Faculty Who Participate in the Point of Care Testing
Number analyzed (Participants) | 15
Number analyzed (survey responses) | 82
laboratories | 1

6. Secondary Outcome: Program Usability
Description: Self report of program usability using the Intervention Usability Scale. Scale values: 1 (strongly disagree) to 5 (strongly agree).
Time Frame: four weeks
Population: Based on engagement and participant feedback during the pilot phases of this study, follow-up surveys were minimized to reduce participant burden. This scale was not implemented for participants, and as such, the outcome cannot be reported.
Arm/Group | PSOM Staff, Trainees, or Faculty Who Participate in the Point of Care Testing
Number analyzed (Participants) | 0

7. Secondary Outcome: User Burden
Description: self report of user burden using the User Burden Scale. Scale values: 0 (not at all) to 5 (extremely).
Time Frame: four weeks
Population: as for outcome 6
Arm/Group | PSOM Staff, Trainees, or Faculty Who Participate in the Point of Care Testing
Number analyzed (Participants) | 0

8. Secondary Outcome: Participant Experience
Description: self report of participant's experience in program using open ended qualitative questions
Time Frame: four weeks
Population: Based on engagement and participant feedback during this study, follow-up questions were minimized to reduce participant burden. Participants had the opportunity to informally share qualitative feedback over the course of the study, but there was not a formal evaluation of participant experience at four weeks. As such, this outcome cannot be reported.
Arm/Group | PSOM Staff, Trainees, or Faculty Who Participate in the Point of Care Testing
Number analyzed (Participants) | 0

9. Secondary Outcome: Program Ease
Description: self report of ease of program using open ended qualitative questions
Time Frame: four weeks
Population: Based on engagement and participant feedback during the pilot phases of this study, follow-up questions were minimized to reduce participant burden. Qualitative interviews were not implemented with participants, and as such, this outcome cannot be reported.
Arm/Group | PSOM Staff, Trainees, or Faculty Who Participate in the Point of Care Testing
Number analyzed (Participants) | 0

10. Secondary Outcome: Program Continuation
Description: self report of interest in program continuing using a Likert Scale. Scale values: 1 (strongly disagree) to 5 (strongly agree).
Time Frame: four weeks
Population: as for outcome 6
Arm/Group | PSOM Staff, Trainees, or Faculty Who Participate in the Point of Care Testing
Number analyzed (Participants) | 0

11. Secondary Outcome: Program Availability
Description: self report of interest in program being more widely available using a Likert Scale. Scale values: 1 (strongly disagree) to 5 (strongly agree).
Time Frame: four weeks
Population: as for outcome 6
Arm/Group | PSOM Staff, Trainees, or Faculty Who Participate in the Point of Care Testing
Number analyzed (Participants) | 0

12. Secondary Outcome: Participant Perspective of Program Implementation and Change in Behavior or Decision-making Process
Description: self report of perspectives of program implementation and change in behavior or decision-making using qualitative open ended questions
Time Frame: one time interview after four weeks of intervention
Population: Based on engagement and participant feedback during this study, follow-up qualitative interviews were not conducted. As such, this outcome cannot be reported.
Arm/Group | PSOM Staff, Trainees, or Faculty Who Participate in the Point of Care Testing
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Fourteen weeks
Arm/Group | PSOM Staff, Trainees, or Faculty Who Participate in the Point of Care Testing
All-Cause Mortality (participants affected / at risk) | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61
Other Adverse Events (participants affected / at risk) | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT05216627/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT05216627/ICF_001.pdf